CLINICAL TRIAL: NCT04629846
Title: A Randomized, Multicenter, Double-Blind, Parallel-Controlled, Phase III Clinical Study to Evaluate QL1209/Pertuzumab in Combination With Docetaxel in Patients With Early-Stage or Locally Advanced HER2-Positive and ER/PR-negative Breast Cancer.
Brief Title: Study in Participants With Early-Stage or Locally Advanced Human Epidermal Growth Factor Receptor (HER) 2-Positive and Estrogen Receptor/Progesterone Receptor Negative Breast Cancer to Evaluate the Efficiency and Safety of Treatment With Trastuzumab Plus (+) QL1209/Pertuzumab + Docetaxel.
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Qilu Pharmaceutical Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: QL1209-301
Record Dates: First submitted 2020-10-28; First posted 2020-11-16 (Actual); Last update posted 2024-04-19 (Actual); Status verified 2024-04

CONDITIONS: Breast Cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — Trastuzumab; pertuzumab; Docetaxel; Surgical Procedures, Operative

STUDY DESIGN:
Intervention Model Description: Parallel Assignment
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Trastuzumab Plus（+） QL1209 + Docetaxel (Experimental): Prior to surgery: trastuzumab, QL1209, and docetaxel for 4 cycles (1 cycle = 21 days) Drug: Docetaxel Drug: QL1209 Drug: Trastuzumab Procedure: Surgery
  Interventions: Drug: Trastuzumab; Drug: QL1209; Drug: Docetaxel; Procedure: surgery
- Trastuzumab Plus（+） Pertuzumab + Docetaxel (Active Comparator): Prior to surgery: trastuzumab,pertuzumab , and docetaxel for 4 cycles (1 cycle = 21 days) Drug: Docetaxel Drug: Pertuzumab Drug: Trastuzumab Procedure: Surgery
  Interventions: Drug: Trastuzumab; Drug: Pertuzumab; Drug: Docetaxel; Procedure: surgery

INTERVENTIONS:
Drug: Trastuzumab — Trastuzumab IV infusion in 3-week cycles. Neoadjuvant treatment: 8 milligrams per kilogram (mg/kg) loading dose for Cycle 1, followed by 6 mg/kg for Cycles 2-4.
  Other Names: Herceptin®
Drug: QL1209 — QL1209 IV infusion in 3-week cycles. Prior to surgery (neoadjuvant treatment): 840 milligrams (mg) loading dose for Cycle 1, followed by 420 mg for Cycles 2-4.
  Other Names: Recombinant anti-HER-2 domain Ⅱ humanized monoclonal antibody injection
  Arms: Trastuzumab Plus（+） QL1209 + Docetaxel
Drug: Pertuzumab — Pertuzumab IV infusion in 3-week cycles. Prior to surgery (neoadjuvant treatment): 840 milligrams (mg) loading dose for Cycle 1, followed by 420 mg for Cycles 2-4.
  Other Names: Perjeta®
  Arms: Trastuzumab Plus（+） Pertuzumab + Docetaxel
Drug: Docetaxel — Docetaxel IV infusion in 3-week cycles. Neoadjuvant treatment: 75 mg/m2 for Cycles 1-4
  Other Names: Docetaxel injection
Procedure: surgery — All participants who are eligible for surgery will undergo surgery and have their pathologic response evaluated.

SUMMARY:
This is a randomized, double-blind, multicenter trial，parallel control designed to evaluate treatment with trastuzumab + QL1209 + docetaxel compared with trastuzumab + pertuzumab + docetaxel in the participants with early-stage or locally advanced HER2-positive and estrogen receptor/progesterone receptor negative breast cancer. The anticipated treatment duration is approximately 140 days.

DETAILED DESCRIPTION:
This is A multi-center, randomized, double-blind, parallel control，comparative clinical trial.

The primary objective is to evaluate whether the clinical efficacy of QL1209 and pertuzumab are similar in patients with early-stage or locally advanced HER2-positive and estrogen receptor/progesterone receptor negative breast cancer.

The secondary objective are to evaluate whether the clinical safety and immunogenicity of QL1209 and pertuzumab are similar in patients with early-stage or locally advanced HER2-positive and estrogen receptor/progesterone receptor negative breast cancer.

ELIGIBILITY:
Inclusion Criteria:

1. Volunteer to participate in this clinical study; Completely understand and know this study as well as sign the informed consent form (ICF);
2. Age ≥ 18 years and ≤ 80 years when ICF is signed;
3. Histologically confirmed invasive breast carcinoma with a primary tumor size of more than (>) 2 centimeters (cm) by standard local assessment technique; Breast cancer stage at presentation: early-stage (T2-3, N0-1, M0) or locally advanced (T2-3, N2 or N3, M0; T4, any N, M0); HER2-positive breast cancer confirmed by immunohistochemistry or HER2 gene amplification by in situ hybridization; Estrogen receptor and Progesterone receptor negative.
4. Eastern Cooperative Oncology Group Performance Status equal to or less than (<=) 1.
5. Baseline left ventricular ejection fracture >= 55% measured by echocardiography (preferred) or multiple gated acquisition scan

Exclusion Criteria:

1. Stage IV metastatic breast cancer;
2. Inflammatory breast cancer;
3. Previous anti-cancer therapy or radiotherapy for any malignancy;
4. History of malignancies other than colorectal cancer within 5 years prior to randomization, excluding cutaneous basal cell carcinoma, cervical carcinoma in situ, and thyroid papillary adenocarcinoma of non-melanoma after radical treatment;
5. Concurrent anti-cancer treatment in another investigational trial, including hormone therapy, bisphosphonate therapy, or immunotherapy;
6. Major surgical procedure within 4 weeks prior to randomization or from which the participant has not fully recovered;
7. Serious cardiac illness or medical condition;
8. Other concurrent serious diseases that may interfere with planned treatment, including severe pulmonary conditions/illness;
9. Sensitivity to any of the study medications, any of the ingredients or excipients of these medications, or benzyl alcohol;
10. Pregnant or lactating

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 517 (Actual)
Dates: Start 2020-11-23 (Actual); Primary Completion 2022-08-22 (Actual); Study Completion 2023-10-24 (Actual)

PRIMARY OUTCOMES:
Total pathologic complete response (tpCR) rate | Approximately 26 months after randomization of the first patient, when all patients have completed the treatment completion/discontinuation visit
  Total pathologic complete response (tpCR) rate, defined as ypT0/is, ypN0 as assessed by an Independent Review Committee (IRC)

SECONDARY OUTCOMES:
Percentage of Participants With tpCR as Assessed by the Local Pathologist | At surgery
  This tpCR was assessed by the local pathologist. tpCR is defined as the absence of any residual invasive cancer on hematoxylin and eosin evaluation of the resected breast specimen and all sampled ipsilateral lymph nodes after completion of neoadjuvant therapy and surgery (that is, ypT0/is, ypN0, in accordance with the current American Joint Committee on Cancer [AJCC] staging system).
Percentage of Participants With Breast Pathologic Complete Response (bpCR) assessed by the IRC | Approximately 26 months after randomization of the first patient, when all patients have completed the treatment completion/discontinuation visit
  This bpCR was assessed by the IRC. bpCR is defined as the absence of any residual invasive cancer on the hematoxylin and eosin evaluation of the resected breast specimen after completion of neoadjuvant therapy and surgery (that is, ypT0/is, in accordance with current AJCC staging system).
Percentage of Participants With bpCR as Assessed by the Local Pathologist | At surgery
  This bpCR was assessed by the local pathologist. bpCR is defined as the absence of any residual invasive cancer on the hematoxylin and eosin evaluation of the resected breast specimen after completion of neoadjuvant therapy and surgery (that is, ypT0/is in accordance with current AJCC staging system).
Percentage of Participants With an Objective Response | Before surgery
  An objective response was defined as the percentage of participants who achieved a complete response or partial response as the best tumor response during the neoadjuvant period (that is, during Cycles 1-4 prior to surgery), as determined by the investigator on the basis of Response Evaluation Criteria in Solid Tumors (RECIST) version 1.1. No confirmation was required for objective response. Only participants with measurable disease at baseline were included in the analysis. The duration of one treatment cycle is 21 days; the administration of therapy in Cycle 5 should not occur until 2 weeks after surgery.

CONTACTS AND LOCATIONS:
Overall Officials: Zhimin Shao, Professor, Principal Investigator — Fudan University; Jin Zhang, Professor, Principal Investigator — Tianjin Medical University Cancer Institute and Hospital
Locations (2):
- China (2):
  - Fudan University Cancer Hospital, Shanghai, Shanghai Municipality
  - Tianjin Medical University Cancer Institution & Hospital, Tianjin, Tianjin Municipality

REFERENCES:
- [Derived] Zuo W, Wang Z, Qian J, Ma X, Niu Z, Ou J, Mo Q, Sun J, Li X, Wang Q, Yao Y, Yu G, Li H, Chen D, Zhang H, Geng C, Qiao G, Zhao M, Zhang B, Kang X, Zhang J, Shao Z. QL1209 (pertuzumab biosimilar) versus reference pertuzumab plus trastuzumab and docetaxel in neoadjuvant treatment for HER2-positive, ER/PR-negative, early or locally advanced breast cancer: A multicenter, randomized, double-blinded, parallel-controlled, phase III equivalence trial. Br J Cancer. 2024 Sep;131(4):668-675. doi: 10.1038/s41416-024-02751-2. Epub 2024 Jun 21. PMID 38906970